CLINICAL TRIAL: NCT06039215
Title: Paramedical Protocol for Ventilation in Acute Respiratory Distress Syndrome: Prospective, Multicenter, Randomized, Controlled, Open-label, Phase III, Cluster Trial With Sequential Permutation
Brief Title: Paramedical Protocol for Ventilation in Acute Respiratory Distress Syndrome
Acronym: PARAVENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APHP191098; 2022-A02716-37 (Other: N° IDRCB)
Record Dates: First submitted 2023-07-12; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome; ARDS; Paramedical care protocol; Mortality
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized, controlled, open-label, phase III, stepped wedge cluster randomized design. This experimental design involves the sequential implementation of an intervention in the clusters included over several periods. The order in which the clusters received the intervention was determined by drawing lots; at the end of the study, all the clusters received the intervention at some point and were observed during a pre- and post-intervention control period (each cluster "is its own control").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Respirator settings are adjusted by nurses according to a pre-established care protocol that complies with international recommendations. The nurse assesses the patient's respiratory status and readjusts the artificial respirator settings if necessary, at least twice a day.
  Interventions: Other: Ventilatory adjustments by nurses
- Control group (No Intervention): The ventilator settings are adjusted in line with the centre's usual practice. No change from usual management of acute respiratory distress syndrome.

INTERVENTIONS:
Other: Ventilatory adjustments by nurses — Respirator settings are adjusted by nurses according to a pre-established care protocol that complies with international recommendations. The nurse assesses the patient's respiratory status and readjusts the artificial respirator settings if necessary, at least twice a day.
  Other Names: Post-intervention period
  Arms: Experimental group

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a frequent pathology in intensive care (around 10% of patients admitted to intensive care and almost a quarter of patients on mechanical ventilation) and a serious one, with a hospital mortality rate of 40%. The main measures that have an effect on mortality in ARDS involve adjustments to the ventilator, known as protective ventilation. In the most severe patients, adjuvant measures such as prone positioning and the use of curarisation in the initial phase of the disease can improve survival. All these measures have been included in the latest national and international recommendations. However, a vast observational study carried out in 50 countries revealed low compliance with these recommendations. More than a third of patients did not receive protective ventilation, and the majority did not receive prone positioning when this was indicated. During weaning from artificial ventilation, it has been widely demonstrated that replacing clinician judgement with the implementation of paramedical care protocols improved weaning and significantly reduced the duration of artificial ventilation. Therefore, investigators hypothesize that the implementation of a paramedical care protocol for ventilation in the acute phase of ARDS improves compliance with recommendations and thus reduces mortality and the duration of artificial ventilation. However, implementation of such a protocol requires operational training for all the nurses in the participating departments. Simulation appears to be the training method of choice, as it is a teaching technique that enables technical and non-technical skills to be passed on with good retention of what has been learnt, as well as assessing what has been learnt. To make it possible to train several dozen nurses within a tight timescale, a partially dematerialized simulation model incorporating innovative e-learning tools will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Intensive care hospitalization;
* Intubation with artificial ventilation;
* ARDS evolving for less than 72 hours. ARDS criteria according to the Berlin definition, as follows:

  * Exposure to a risk factor for ARDS or onset/aggravation of pulmonary symptoms within the previous 7 days ;
  * Respiratory distress not fully explained by cardiac failure or volume overload, with exclusion of hydrostatic edema in the absence of exposure to a risk factor for ARDS;
  * Hypoxemia with PaO2/FiO2 ratio < 300 mm Hg under PEEP ≥ 5 cmH2O ;
  * Bilateral opacities on chest X-ray, lung ultrasound or chest CT, not fully explained by pleural effusions, atelectasis or nodules.
* Blood pressure monitoring
* Affiliation to the social security system.
* Written informed consent (patient, relative) or inclusion in emergency situation.

Exclusion Criteria:

* Long-term oxygen therapy;
* Pneumothorax or drained pleurisy;
* Documented pulmonary embolism;
* Intracranial hypertension;
* ARDS refractory to inclusion, i.e.: i) oxygen partial pressure on inspired oxygen fraction a ratio (PaO2/FiO2) <80 mm Hg or plateau pressure (Pplat) > 32 cmH2O despite optimization of mechanical ventilation (tidal volume (Vt) set at 6 mL/kg weight predicted by height, FiO2 ≥80% and positive expiratory pressure (PEEP) ≥10 cmH2O) and despite the use of complementary therapies (including prone and/or inhaled nitric oxide); or ii) pH <7. 25 with PaCO2 ≥60 mm Hg;
* ARDS evolving for more than 72 hours with intubation and mechanical ventilation;
* Patient deprived of liberty;
* Patient under legal protection (guardianship or curatorship);
* Known pregnancy or breast-feeding (a pregnancy test will be performed prior to inclusion in patients of childbearing age).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Mortality rate and number of days without mechanical ventilation | 28 days
  The primary endpoint will be a combination of mortality and the number of days without mechanical ventilation at D28. This composite criterion will be prioritised so that survival is given priority in the analysis over the shorter duration of mechanical ventilation.

SECONDARY OUTCOMES:
Mesure of tidal volume ventilation | Up to Day 7
Mesure of plateau pressure | Up to Day 7
Mesure of positive end-expiratory pressure (PEEP) | Up to Day 7
Mesure of FiO2 | Up to Day 7
Oxygenation | Up to Day 7
  arterial blood gases and SpO2
Number of days without mechanical ventilation | Up to Day 28
Number of days without catecholamine | Up to Day 28
Number of days without continuous sedation | Up to Day 28
Duration of mechanical ventilation . | Up to Day 28
  from intubation to successful extubation
Occurrence of mechanically ventilated pneumothorax | Up to Day 28
Duration of Acute respiratory distress syndrome | UP to Day 28
  defined as the day on which the 1st test of spontaneous ventilation was performed
Duration of weaning from mechanical ventilation | Up to Day 28
  measured as the time between the 1st test of spontaneous ventilation and successful extubation (patient alive and without reintubation within 7 days of extubation).
Number of participants with rescue therapy | Up to Day 28
Rate of re-intubation | Up to Day 28
Rate of use of non-invasive ventilation and curative high-flow oxygen therapy | Up to Day 28
Tracheostomy rate | Up to Day 28
Length of stay in intensive care and in hospital. | Up to day 28
Number of deaths in ICU and hospital | Up to Day 28
Number of nurses trained in paramedical protocol per center. | Up to 26 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique-Hôpitaux de Paris service de santé publique, Créteil, Creteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION